CLINICAL TRIAL: NCT01671319
Title: Phase II Study of Dose-Dense TC (Docetaxel + Cyclophosphamide) With Pegfilgrastim Support for Adjuvant Therapy of pN0, pN1 or Nx Breast Cancer
Brief Title: Dose Dense TC + Pegfilgrastim Support for Breast Cancer
Acronym: ddTC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CO10104; 2011-0062 (Other: Institutional Review Board); NCI-2011-03640 (Registry Identifier: NCI Trial ID); A535900 (Other: UW Madison); SMPH\ONCOLOGY\ONCOLOGY (Other: UW Madison)
Record Dates: First submitted 2011-08-05; First posted 2012-08-23 (Estimated); Results first posted 2017-10-12 (Actual); Last update posted 2019-11-27 (Actual); Status verified 2017-09

CONDITIONS: Female Breast Cancer
Keywords: breast cancer; female; women; adjuvant
MeSH Terms: conditions — Breast Neoplasms | interventions — Docetaxel; Cyclophosphamide; pegfilgrastim

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- dose dense TC + pegfilgrastim (Experimental): Docetaxel + Cyclophosphamide chemotherapy given every 2 weeks x 4 cycles plus pegfilgrastim given 24-48 hours post day 1 of each cycle
  Interventions: Drug: docetaxel + cyclophosphamide + pegfilgrastim

INTERVENTIONS:
Drug: docetaxel + cyclophosphamide + pegfilgrastim — docetaxel 75 mg/m2 + cyclophosphamide 600 mg/m2 IV every 2 weeks x 4 cycles plus pegfilgrastim 6mg sq 24-48 hours post day 1 of each cycle
  Other Names: Taxotere, Cytoxan, Neulasta

SUMMARY:
The purpose of this study is to determine the feasibility of giving standard TC chemotherapy on a dose dense schedule (ddTC) as well as evaluating the nature and frequency of ddTC side effects.

DETAILED DESCRIPTION:
A standard chemotherapy treatment option for breast cancer after surgery (adjuvant therapy) is docetaxel + cyclophosphamide (TC). This study looks at a different schedule for giving the same adjuvant chemotherapy so that treatment can be completed faster (in 8 weeks rather than 12 weeks). This study uses a growth factor drug, pegfilgrastim, to help build blood cells that are lowered because of chemotherapy, making it possible to receive TC treatment every 2 weeks (referred to as "dose dense TC" or "ddTC") instead of the standard 3 week schedule. The main study procedures are blood draws, chemotherapy treatment, physical exams, and pegfilgrastim injections.

ELIGIBILITY:
Inclusion Criteria:

* histologically confirmed invasive carcinoma of the female breast, status post definitive surgery (lumpectomy or mastectomy plus nodal evaluation if feasible). Patients must initiate therapy with ddTC within 84 days of the last breast or axillary surgery performed for curative intent
* candidate for chemotherapy by the treating oncologist
* Patients with pN2 or pN3 disease are NOT explicitly excluded. However, patients with N2 or N3 disease MUST be reviewed with the PI or study chair before being enrolled on the study as TC would not normally be considered adequate therapy for such patients.
* Patients with bilateral, synchronous invasive breast cancer are eligible as long as both primary tumors meet the eligibility criteria.
* Patients with estrogen-receptor (ER) and/or progesterone receptor (PR) negative, positive, or unknown tumors are eligible.
* Patients with HER2 positive, negative or unknown disease are eligible for this trial. Patients whose tumors are HER2 positive by either immunohistochemistry (IHC) 3+ staining or demonstrate gene amplification by FISH should receive trastuzumab, following completion of adjuvant cytotoxic therapy with 4 cycles of ddTC.
* There must be negative surgical margins for invasive cancer and DCIS. LCIS is acceptable at the margin.
* Patients with multi-centric breast cancer are eligible as long as all known disease is resected from the breast with negative margins.
* Age >18 years.
* ECOG performance status ≤ 1
* Women of childbearing potential should have a negative urine or blood beta-HCG, and must agree to contraception if engaging in sexual activity. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately. Women must not be pregnant or nursing as the chemotherapy drugs used in this study may cause harm to a fetus or newborn.
* Ability to understand and the willingness to sign a written informed consent document.
* Platelets >/=100,000/μl within 4 weeks of registration.
* Absolute neutrophil count (ANC) >/= 1,500/μl within 4 weeks of registration.
* Total bilirubin within normal institutional limits within 4 weeks of registration.
* Alkaline phosphatase (alk phos) ≤ 2.5 X institutional Upper Limit of Normal (ULN) within 4 weeks of registration.
* AST (SGOT)/ALT(SGPT) ≤ 1.5X ULN
* Creatinine within normal institutional limits OR Creatinine clearance>/= 60 mL/min/1.73 m2 for patients with creatinine levels above normal
* If patient has received tamoxifen or another selective estrogen receptor modulator (SERM) for prevention or for other indications (not for treatment of this cancer), they have been discontinued prior to enrollment.

Exclusion Criteria:

* Patient has received previous trastuzumab, chemotherapy, hormonal therapy, or other anti-cancer agents (including investigational agents) for this malignancy.
* Patient will be receiving GNRH agonists such as goserelin (Zoladex) or leuprolide acetate (Lupron) concomitantly with chemotherapy for the purpose of preventing breast cancer recurrence.
* Patient has inflammatory breast cancer (pT4d) or metastatic breast cancer.
* Patient has uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia or psychiatric illness/social situations that would limit compliance with study requirements.
* Patient has pre-existing persistent neuropathy.
* The patient has received prior chemotherapy or radiotherapy or any malignancy within the past 2 years.
* Patient has received prior docetaxel or cyclophosphamide within the past 5 years.
* Patient has known contraindication or hypersensitivity to docetaxel, cyclophosphamide or pegfilgrastim.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2011-06; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amye J Tevaarwerk, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin Carbone Cancer Center, Madison, Wisconsin, United States

REFERENCES:
- [Result] Burkard ME, Wisinski KB, Njiaju UO, Donohue S, Hegeman R, Stella A, Mansky P, Shah V, Goggins T, Qamar R, Dietrich L, Kim K, Traynor AM, Tevaarwerk AJ. Feasibility of 4 cycles of docetaxel and cyclophosphamide every 14 days as an adjuvant regimen for breast cancer: a Wisconsin Oncology Network study. Clin Breast Cancer. 2014 Jun;14(3):205-11. doi: 10.1016/j.clbc.2013.10.018. Epub 2013 Oct 26. PMID 24342730
- See also: University of Wisconsin Carbone Cancer Center — https://cancer.wisc.edu/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was performed through the Wisconsin Oncology Network, a regional oncology network, at a combination of academic and community practice sites. Patients were enrolled between June 2011 and June 2012.
Period: Overall Study
Arm/Group | Dose Dense TC + Pegfilgrastim
Started | 42
Completed | 41
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: Women with early stage breast cancer.
Arm/Group | Dose Dense TC + Pegfilgrastim
Number analyzed (Participants) | 41
Age, Continuous [Median (Full Range); unit: years] | 54 [28 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 39
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 41
Pre- vs. Postmenopausal [Count of Participants; unit: Participants]
  Premenopausal | 15
  Postmenopausal | 26
Staging Criteria [Count of Participants; unit: Participants] — Participants were staged according to the American Joint Committee on Cancer (AJCC) staging manual.
  Node-negative: cancer has not spread to the lymph nodes Node-positive: cancer that has spread to the lymph nodes T1 and T2 refer to the size and/or extent of the main tumor. The higher the number after the T, the larger the tumor or the more it has grown into nearby tissues.
  Participants
    Node-negative | 30
    Node-positive | 10
    Nodes unknown | 1
    T1 | 21
    T2 | 20
Receptor Status [Count of Participants; unit: Participants]
  Hormone receptor-postive | 29
  HER2-positive | 1
  Triple negative | 11
Final Surgery [Count of Participants; unit: Participants]
  Mastectomy | 20
  Breast conservation | 21

OUTCOME MEASURES:

1. Primary Outcome: Feasibility for Dose-dense TC Therapy: Number of Participants Receiving at Least 90% of Total Dose of Therapy
Description: Evaluate feasibility of delivering 4 cycles (1 cycle = 2 weeks) of docetaxel and cyclophosphamide (TC) on a dose-dense (q2week) schedule with pegfilgrastim support. This regimen will be referred to as dose-dense (dd)TC. Feasibility defined by at least 60% of patients receiving 90% of the total dose of therapy within 10 weeks.
Time Frame: 4 cycles each 2 weeks in length for a total of 8 weeks, up to 10 weeks
Population: Of 42 participants, 41 were evaluable for outcome measure analysis.
Measure: Number; unit: participants
Arm/Group | Dose Dense TC + Pegfilgrastim
Number analyzed (Participants) | 41
participants | 37

2. Secondary Outcome: Incidence of Febrile Neutropenia
Description: Neutropenic fever was anticipated to be a clinically significant toxicity that would limit the maximal density of TC therapy.
Time Frame: Up to 10 weeks
Population: Of 42 participants, 41 were evaluable for outcome measure analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Dense TC + Pegfilgrastim
Number analyzed (Participants) | 41
Participants | 1

3. Secondary Outcome: Incidence of Neuropathy
Description: Neuropathy was anticipated to be a clinically significant toxicity that would limit the maximal density of TC therapy.
Time Frame: Up to 10 weeks
Population: Of 42 participants, 41 were evaluable for outcome measure analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Dense TC + Pegfilgrastim
Number analyzed (Participants) | 41
Participants
  Sensory neuropathy | 5
  Motor neuropathy | 1
  No incidence of neuropathy | 35

ADVERSE EVENTS:
Description: Toxicity assessments were made one day 1 of each cycle, and as indicated clinically.
Arm/Group | Dose Dense TC + Pegfilgrastim
Serious Adverse Events (participants affected / at risk) | 4/42
Other Adverse Events (participants affected / at risk) | 42/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Dense TC + Pegfilgrastim (N=42)
Febrile neutropenia (Infections and infestations) | 1 (1)
Perforation, GI (Gastrointestinal disorders) | 1 (1)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Dense TC + Pegfilgrastim (N=42)
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 6 (11)
Alkaline phosphatase (Metabolism and nutrition disorders) | 9 (10)
Allergic reaction/hypersensitivity (including drug fever) (Immune system disorders) | 3 (3)
Allergic rhinitis (including sneezing, nasal stuffiness, postnasal drip) (Immune system disorders) | 2 (2)
ALT, SGPT (serum glutamic pyruvic transaminase) (Metabolism and nutrition disorders) | 16 (20)
Anorexia (Gastrointestinal disorders) | 11 (13)
Arthritis (non-septic) (Musculoskeletal and connective tissue disorders) | 1 (1)
AST, SGOT(serum glutamic oxaloacetic transaminase) (Metabolism and nutrition disorders) | 9 (11)
Auditory/Ear - Ear pain (Ear and labyrinth disorders) | 1 (1)
Autoimmune reaction (Immune system disorders) | 1 (1)
Bilirubin (hyperbilirubinemia) (Metabolism and nutrition disorders) | 2 (2)
Bruising (in absence of Grade 3 or 4 thrombocytopenia) (Skin and subcutaneous tissue disorders) | 1 (1)
Calcium, serum-high (hypercalcemia) (Metabolism and nutrition disorders) | 2 (3)
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 13 (13)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Creatinine (Metabolism and nutrition disorders) | 5 (5)
Cytokine release syndrome/acute infusion reaction (Immune system disorders) | 1 (1)
Dehydration (Gastrointestinal disorders) | 2 (2)
Dermatology/Skin (Skin and subcutaneous tissue disorders) | 8 (9)
Diarrhea (Gastrointestinal disorders) | 14 (21)
Distension/bloating, abdominal (Gastrointestinal disorders) | 2 (2)
Dizziness (Nervous system disorders) | 4 (4)
Dry eye syndrome (Eye disorders) | 2 (3)
Dry mouth/salivary gland (xerostomia) (Gastrointestinal disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 6 (7)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Edema: limb (Endocrine disorders) | 6 (6)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 34 (71)
Febrile neutropenia (Infections and infestations) | 2 (2)
Fever (General disorders) | 4 (4)
Flushing (Skin and subcutaneous tissue disorders) | 4 (4)
Gastritis (including bile reflux gastritis) (Gastrointestinal disorders) | 1 (1)
Gastrointestinal (Gastrointestinal disorders) | 3 (4)
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 14 (32)
Hair loss/alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 21 (26)
Heartburn/dyspepsia (Gastrointestinal disorders) | 5 (6)
Hemoglobin (Blood and lymphatic system disorders) | 32 (59)
Hemorrhage, pulmonary/upper respiratory - Nose (Blood and lymphatic system disorders) | 2 (3)
Hemorrhage/Bleeding (Blood and lymphatic system disorders) | 2 (3)
Hot flashes/flushes (Endocrine disorders) | 4 (5)
Hypothermia (General disorders) | 1 (1)
Infection (Infections and infestations) | 8 (9)
Injection site reaction/extravasation changes (General disorders) | 6 (9)
Insomnia (General disorders) | 5 (5)
Irregular menses (change from baseline) (Reproductive system and breast disorders) | 1 (1)
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 4 (4)
Lymphopenia (Blood and lymphatic system disorders) | 1 (1)
Mood alteration - Anxiety (Nervous system disorders) | 4 (5)
Mucositis/stomatitis (clinical exam) - Oral cavity (Gastrointestinal disorders) | 17 (21)
Muscle weakness, generalized or specific area (not due to neuropathy) - Extremity-lower (Musculoskeletal and connective tissue disorders) | 1 (1)
Nail changes (Skin and subcutaneous tissue disorders) | 16 (17)
Nasal cavity/paranasal sinus reactions (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Nausea (Gastrointestinal disorders) | 18 (29)
Neurology - Other (Nervous system disorders) | 4 (4)
Neuropathy: motor (Nervous system disorders) | 1 (1)
Neuropathy: sensory (Nervous system disorders) | 22 (30)
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 4 (5)
Ocular/Visual - Itchy eyes (Eye disorders) | 2 (2)
Pain (General disorders) | 33 (77)
Palpitations (Cardiac disorders) | 1 (1)
Perforation, GI - Colon (Gastrointestinal disorders) | 1 (1)
Phlebitis (including superficial thrombosis) (Vascular disorders) | 1 (1)
Phosphate, serum-low (hypophosphatemia) (Metabolism and nutrition disorders) | 1 (1)
Photosensitivity (Skin and subcutaneous tissue disorders) | 2 (2)
Platelets (Blood and lymphatic system disorders) | 11 (15)
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 1 (1)
Pulmonary/Upper Respiratory - Other (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 8 (14)
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 6 (7)
Rash: erythema multiforme (e.g., Stevens-Johnson syndrome, toxic epidermal necrolysis) (Skin and subcutaneous tissue disorders) | 4 (5)
Rash: hand-foot skin reaction (Skin and subcutaneous tissue disorders) | 12 (14)
Renal/Genitourinary - Dysuria (Renal and urinary disorders) | 1 (1)
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 3 (4)
Supraventricular and nodal arrhythmia - Sinus bradycardia (Cardiac disorders) | 1 (1)
Supraventricular and nodal arrhythmia - Sinus tachycardia (Cardiac disorders) | 2 (2)
Sweating (diaphoresis) (General disorders) | 1 (1)
Taste alteration (dysgeusia) (Gastrointestinal disorders) | 11 (12)
Tremor (Nervous system disorders) | 1 (1)
Urinary frequency/urgency (Renal and urinary disorders) | 1 (1)
Vaginal mucositis (Reproductive system and breast disorders) | 1 (1)
Vision-blurred vision (Eye disorders) | 1 (1)
Voice changes/dysarthria (e.g., hoarseness, loss or alteration in voice, laryngitis) (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Vomiting (Gastrointestinal disorders) | 2 (3)
Watery eye (epiphora, tearing) (Eye disorders) | 15 (16)
Weight gain (General disorders) | 1 (1)
Weight loss (General disorders) | 1 (1)
Wound complication, non-infectious (Skin and subcutaneous tissue disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No